CLINICAL TRIAL: NCT00291278
Title: The Effects of Endometriosis on Bone Mineral Density
Brief Title: Effects of Endometriosis on Bone Mineral Density
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060091; 06-CH-0091
Record Dates: First submitted 2006-02-11; First posted 2006-02-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; Bone Mineral Density; Osteopenia; Osteoporosis; DEXA Scan; Menopause; Screening; Healthy Volunteer; HV
MeSH Terms: conditions — Endometriosis; Bone Diseases, Metabolic; Osteoporosis

SUMMARY:
This study will compare bone mass in women with a history of endometriosis, a disease in which the lining of the uterus grows on nearby tissues, to that of women who have not had endometriosis. Endometriosis may be treated with medication or surgery, or both. Because uterine tissue grows more when estrogen levels are high, medical treatment is designed to lower estrogen. Decreased estrogen, however, is often associated with weak bones and hot flashes. Also, women with endometriosis may have lower bone density as a consequence of their disease. This study will look at bone density in these women, particularly to see if areas other than the lower back may be affected.

Regularly menstruating women between 40 and 50 years old, with or without a history of endometriosis, may be eligible for this study. Candidates are screened by telephone; women with endometriosis are asked to provide documentation of their endometriosis before beginning the study.

Study participants undergo the following tests and procedures:

* Medical history and blood sample collection
* Questionnaires about exercise activity, calcium intake, menstrual cycle history, cigarette use and medication history
* DEXA scan: This test evaluates the strength of the bones in the back, wrist, and hip. The DEXA scanner uses low-energy x-rays to determine bone density. Scans are done of the lower spine, upper thigh, hip, and the entire body. For the test, the subject lies on the scanning table. Each scan takes about 3 minutes, and the entire procedure may take as long as 1 hour.

DETAILED DESCRIPTION:
After peaking in the third decade, bone mineral density (BMD) decreases slowly over time, with a more dramatic short-term decline at the time of menopause. Because of the association with osteoporosis and fracture, evaluation of BMD at the time of menopause is recommended, as is identification and treatment of any reversible causes of bone mineral loss. Most studies of women with endometriosis have shown no change or decreased BMD, while rats with induced endometriosis had a marked decrease in BMD. Often, studies in women did not control for factors that are known to affect bone density such as body mass index (BMI), exercise, or calcium intake. To address the question of whether endometriosis is associated with a change in BMD, we previously matched healthy volunteers and endometriosis patients for age, race, BMI, exercise level and calcium intake and compared BMD in the two groups. We found a decrease in BMD in women aged 40 - 50 who had a history of endometriosis, in comparison to women who did not have such a history. This study will expand that experience by studying more women aged 40 - 50 years with a history of endometriosis and matching them to women of the same race with similar age and BMI, who do not have a history of endometriosis. Participants will fill out a questionnaire about their medical, exercise and dietary history and will provide a single blood sample. A bone density study will be done and results will be made available to the participants.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Regularly cycling women between the ages of 40 and 50 with surgically documented endometriosis (preferably biopsy proven, but unequivocal operative reports may allow inclusion).

     OR
  2. Regularly cycling women between the ages of 40 and 50 who are healthy volunteers.

Women will be matched by ethnicity, by BMI within 5 kg/M(2), and by age (at the time of DEXA) in two groups: 40 - 45 years and 45 - 50 years.

EXCLUSION CRITERIA:

Women who are pregnant or lactating or who have abnormalities in the medical history or screening laboratory tests that might contribute to abnormal BMD (e.g. hypercalcemia, renal failure) will not be enrolled

We will not include women who currently or have previously taken medications known to affect bone mineral density (e.g. thyroid hormone suppression, supraphysiologic glucocorticoids, GnRH, dilantin) or those that suggest menstrual abnormalities (fertility drugs), but we will consider other prescription drug use on a case-by-case basis.

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2006-02-07; Study Completion 2009-02-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hearns-Stokes RM, Santoro NF, Simon JA. Surgically induced endometriosis attenuates accrual of bone mineral density in growing rats. Am J Obstet Gynecol. 2001 Feb;184(3):331-5. doi: 10.1067/mob.2001.110025. PMID 11228482
- [Background] Lopez-Castejon A, Revilla M, Hernandez ER, Villa LF, Rico H, Cortes J. Effect of induced uterine retroversion on bone mass in rats. Eur J Obstet Gynecol Reprod Biol. 1999 Mar;83(1):101-4. doi: 10.1016/s0301-2115(98)00304-2. PMID 10221617
- [Background] Comite F, Delman M, Hutchinson-Williams K, DeCherney AH, Jensen P. Reduced bone mass in reproductive-aged women with endometriosis. J Clin Endocrinol Metab. 1989 Oct;69(4):837-42. doi: 10.1210/jcem-69-4-837. PMID 2778037